CLINICAL TRIAL: NCT06881095
Title: Immediate Dental Implant Installation With and Without Socket Shield Technique in Aesthetic Zone
Acronym: socket shield
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Islam Ahmed Elsayed, master degree( Principal Investigator), Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: islam123
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Immediate Dental Implants; Thin Labial Plate of Bone Pre-extraction; Hopeless Tooth in Esthetic Zone
Keywords: socket shield technique; partial extraction therapy; immediate dental implant
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: non restorable anterior teeth with thin labial plate of bone
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- socket shield technique group (study group) (Experimental): the socket shield technique group (study group): 10 patients will have immediate implant placement with socket shield technique.
  * conventional immediate dental implant technique (control group): 10 patients will have immediate implant placement with conventional technique without socket shield technique.
  preparation of shield: the root will be sectioned in a mesio-distal direction along its long axis, sectioning divided the tooth root into one facial third and two palatal thirds, Periotomes will then be inserted between the palatal root section and the alveolar socket wall to sever the PDL and this section of root was then carefully delivered so as not to disturb the facial root section, the remaining root section was then reduced coronally to 1 mm above the alveolar crest.
  The tooth socket's palatal wall and apex will be then curetted to remove any tissue or infective remnants and the root section was checked for immobility with a sharp probe.
  After completion of th
  Interventions: Procedure: socket shield technique group (study group)
- conventional immediate implant without socket shield technique(control group) (Experimental): conventional immediate implant without socket shield technique:
  • After administration of local anesthesia, atraumatic tooth extraction by extraction forceps and Periotomes, an osteotomy was then sequentially prepared according to manufacturer instructions and a suitable implant then inserted and placement of cover screw. However, the soft tissue contour formed after healing may need some modification prior to impression taking. Suturing around the healing abutment, suture will be removed one week post surgically and then healing abutment and final prosthetic loading will be done after 4-6 months.
  Interventions: Procedure: conventional immediate implant without socket shield technique

INTERVENTIONS:
Procedure: socket shield technique group (study group) — immediate implant installation with socket shield technique: After administration of local anesthesia, the root will be sectioned in a mesio-distal direction along its long axis, sectioning divided the tooth root into one facial third and two palatal thirds.
  Periotomes will then be inserted between the palatal root section and the alveolar socket wall to sever the PDL and this section of root was then carefully delivered so as not to disturb the facial root section, the remaining root section was then reduced coronally to 1 mm above the alveolar crest.
  The tooth socket's palatal wall and apex will be then curetted to remove any tissue or infective remnants, and the root section was checked for immobility with a sharp probe.
  After completion of the previous steps, the tooth root here will be known as the socket- shield (SS). An osteotomy was then sequentially prepared according to manufacturer
  Other Names: partial extraction therapy
  Arms: socket shield technique group (study group)
Procedure: conventional immediate implant without socket shield technique — • After administration of local anesthesia, atraumatic tooth extraction by extraction forceps and Periotomes, an osteotomy was then sequentially prepared according to manufacturer instructions and a suitable implant then inserted and placement of cover screw. However, the soft tissue contour formed after healing may need some modification prior to impression taking. Suturing around the healing abutment, suture will be removed one week post surgically and then healing abutment and final prosthetic loading will be done after 4-6 months.
  Arms: conventional immediate implant without socket shield technique(control group)

SUMMARY:
20 patients with non-restorable anterior teeth underwent extraction with immediate implant installation using either the immediate implant with socket shield technique or the conventional immediate dental implant.

the socket shield technique group (study group): 10 patients will have immediate implant placement with the socket shield technique.

* conventional immediate dental implant technique (control group): 10 patients will have immediate implant placement with conventional technique.

DETAILED DESCRIPTION:
20 patients with non-restorable anterior teeth underwent extraction with immediate implant installation randomized to two groups immediate dental implant with the socket shield technique group (study group): 10 patients will have immediate implant placement with socket shield technique.

* conventional immediate dental implant technique (control group): 10 patients will have immediate implant placement with conventional technique without socket shield technique.

preparation of shield: the root will be sectioned in a mesio-distal direction along its long axis, sectioning divided the tooth root into one facial third and two palatal thirds, Periotomes will then be inserted between the palatal root section and the alveolar socket wall to sever the PDL and this section of root was then carefully delivered so as not to disturb the facial root section, the remaining root section was then reduced coronally to 1 mm above the alveolar crest.

The tooth socket's palatal wall and apex will be then curetted to remove any tissue or infective remnants and the root section was checked for immobility with a sharp probe.

After completion of the previous steps, the tooth root here will be known as the socket- shield (SS). An osteotomy was then sequentially prepared according to manufacturer instructions and a suitable implant then inserted palatal to the SS.

ELIGIBILITY:
Inclusion Criteria:

- 1. Non restorable maxillary anterior teeth without periapical pathology that may affect the success of dental implants.

2. Interarch space enough for prosthetic rehabilitation. 3. Presence of posterior teeth or prosthesis that maintain occlusal bite. 4. Adult patients. 5. Good oral hygiene.

Exclusion Criteria:

- 1. Edentulous anterior maxillary region. 2. Bad oral hygiene. 3. Patients with any relevant systemic diseases that affect soft tissue or bone healing.

4. Patients with parafunctional habits (bruxism and clenching). 5. Uncooperative patients. 6. Heavy smokers.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-05-12 (Estimated); Study Completion 2025-06-16 (Estimated)

PRIMARY OUTCOMES:
labial bone thickness | 6 months
  1. labial bone thickness measuring thickness of labial bone labial to the implant by (CBCT) Cone beam computed tomography
marginal bone loss | 6 months

SECONDARY OUTCOMES:
bone density around dental implant | 6 months
  bone density around dental implant by Cone beam computed tomography
implant secondary stability | 6 months
  Secondary implant stability: will be recorded just after uncovery using Resonance frequency analysis (RFA) device * (Osstell).
implant success | 6 months
  absence of infection, fistula formation or implant mobility

CONTACTS AND LOCATIONS:
Overall Officials: islam ahmed abo elela, master study, Principal Investigator — faculty of dentistry tanta university; Ibrahim mohammed nowair, professor, Principal Investigator — faculty of dentistry tanta university; Rafic ramadan bedir, professor, Principal Investigator — faculty of dentistry tanta university; Wesam Hamed Elsaadany, lecturer, Principal Investigator — faculty of dentistry tanta university
Locations (1):
- Faculty of Dentistry, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No